CLINICAL TRIAL: NCT02276079
Title: The Effect of Exercise on Neurorecovery Following Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Clinical & Translational Science Institute (Unknown); American Psychological Foundation (Other); American Psychological Association (APA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400882
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Brain Concussion
Keywords: Mild Traumatic Brain Injury; Aerobic Exercise; Brain-Derived Neurotrophic Factor
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mTBI Aerobic Exercise Group (Experimental): Participants are two-three weeks post-mild traumatic brain injury are randomized to receive a daily aerobic exercise intervention lasting 1-week.
  Interventions: Behavioral: Aerobic Exercise
- mTBI Non-Aerobic Exercise Group (Experimental): Participants are two-three weeks post-mild traumatic brain injury are randomized to receive a daily non-aerobic exercise intervention lasting 1-week.
  Interventions: Behavioral: Non-Aerobic Exercise
- Non-injured Reference Group (No Intervention): Non-injured, healthy participants will serve as a reference group for functional outcome measures.

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise will consist of riding a stationary bicycle at moderate intensity for 2 consecutive, 20-minute periods with a 5-minute break in between. Moderate intensity is defined as maintaining 65-75% of estimated maximum heart rate based on the calculation (HRmax = 208 - 0.7 × age).
  Arms: mTBI Aerobic Exercise Group
Behavioral: Non-Aerobic Exercise — Non-Aerobic exercise will consist of very low-intensity movements including static stretching and toning exercises.Participants will complete 2 consecutive, 20-minute periods with a 5-minute break in between, mirroring the aerobic exercise condition. Heart rate will be monitored by research staff to ensure that it remains below 50% of estimated maximum heart rate.
  Arms: mTBI Non-Aerobic Exercise Group

SUMMARY:
The study is a "proof-of-principle" project to examine the safety and feasibility of implementing a 1-week aerobic exercise program in the post-acute phase after mild traumatic brain injury (mTBI). The study will define the extent to which the exercise program improves recovery from mTBI in terms of relevant functional outcomes (cognition, mood, and physical status) and biomarkers (peripheral brain-derived neurotrophic factor [BDNF] concentration).

DETAILED DESCRIPTION:
This is a "proof-of-principle" project for human subjects to examine the safety and feasibility of implementing a 1-week aerobic exercise program in the post-acute phase after mild traumatic brain injury (mTBI). This study will define the extent to which the exercise program improves recovery from mTBI in terms of relevant functional outcomes (cognition, mood, and physical status) and biomarkers (peripheral brain-derived neurotrophic factor [BDNF] concentration). This project will also lay the foundation for understanding the relationship between exercise and BDNF in the area of mTBI neurorecovery, thereby allowing future studies to develop best-practice methods for implementing exercise interventions as a treatment option for brain injuries.

ELIGIBILITY:
Mild traumatic brain injury (mTBI) group:

Inclusion Criteria:

* Meet criteria for mTBI as set forth by the American Congress of Rehabilitation Medicine
* mTBI was sustained 14-25 days before beginning the exercise intervention

Exclusion Criteria:

* comorbid orthopaedic injury that inhibits movement
* history of serious psychiatric disturbance with hospitalization,
* prior history of neurologic disease,
* current or past history of substance abuse disorder,
* diabetes
* previous history of moderate or severe head injury,
* neurological disorder unrelated to TBI (e.g., seizure disorder)
* physician recommendations against exercise
* non-English speakers

Non-injured Group:

Inclusion Criteria:

- Gainesville, Florida community member

Exclusion Criteria:

* History of mTBI or other brain injury in the past year
* comorbid orthopaedic injury that inhibits movement
* history of serious psychiatric disturbance with hospitalization,
* prior history of neurologic disease,
* current or past history of substance abuse disorder,
* diabetes
* previous history of moderate or severe head injury,
* neurological disorder unrelated to TBI (e.g., seizure disorder)
* physician recommendations against exercise
* non-English speakers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Score on the Sport Concussion Assessment Tool (SCAT3) | Baseline and up to day 8
  Obtained from the 22-item symptom evaluation included in the Sport Concussion Assessment Tool (SCAT3). The participant's present experience of each symptom is rated on a likert scale from 0 (none) to 6 (severe). The symptom score represents how many symptoms the participant endorses experiencing at a level greater than 0 (maximum 22 points).
Change in Symptom Severity on the Sport Concussion Assessment Tool (SCAT3) | Baseline and up to day 8
  Symptom evaluation included in the Sport Concussion Assessment Tool (SCAT3). The participant's present experience of each symptom is rated on a likert scale from 0 (none) to 6 (severe). The symptom severity represents the total summed severity ratings for all symptoms (maximum 132 points).
Change in sleep quality | Baseline and up to day 8
  Obtained from the Medical Outcomes Sleep Scale (MOS). This measure has 12 items and asks the participant to rate different aspects of their sleep experiences and sleep quality. The first two questions inquire about sleep times and the remaining questions utilize a likert scale ranging from 1 (all of the time) to 6 (none of the time). Some items are reverse scored and the scale yields several subscale measures, so scoring rules depend on the specific subscale.
Change in postural stability | Baseline and up to day 8
  The Balance Error Scoring System (BESS) will be used to measure postural stability, which is sensitive to deficits in balance following mild head injury. A modified version of (SCAT3) will be used. It includes three different stances, double leg, single leg, and tandem stance. A point is added for committing an error during the test interval and if the participant is unable to maintain his or her balance for more than 5 seconds, the trial is discontinued and maximum points are awarded. The total score ranges from 0 (better postural stability) to 30 (worse postural stability).
Change in verbal learning and memory | Baseline and up to day 8
  Measured by the California Verbal Learning Test, 2nd Edition (CVLT-II). This test measures word recall and assesses the following skills: immediate recall, short delay free recall, short delay cued recall, long delay free recall, long delay cued recall, and long delay recognition.
Change in auditory-linguistic memory | Baseline and up to day 8
  Measured by the Wechsler Memory Scale, 3rd Edition (WMS-III), Logical Memory subtests. Two stories are read to participants and then they are asked to freely recall items after a short and a long delay. A recognition trial is administered following the long delay.
Change in word-fluency | Baseline and up to day 8
  Measured by the Controlled Oral Word Association (COWA). Participants are asked to say as many words beginning with a specified letter as they can in a one minute time period. Three trials with different letters are administered.
Change in semantic fluency | Baseline and up to day 8
  Measured by the Verbal Fluency Test - Categories. Participants are asked to say as many items belonging to a specified semantic category as they can in a one minute time period.
Change in psychomotor/executive functioning | Baseline and up to day 8
  Measured by the Delis-Kaplan Executive Functioning System (D-KEFS), Trail Making Test. The test consists of five different conditions where participants are asked to draw trails according to specified rules.
Change in problem solving and abstract reasoning | Baseline and up to day 8
  Measured by the Wisconsin Card Sorting Test (WCST). Initially, a number of stimulus cards are presented to the participant. The participant is told to match the cards, but not how to match; however, he or she is told whether a particular match is right or wrong. A total of 128 cards are played.
Change in attention | Baseline and up to day 8
  Measured by the Wechsler Adult Intelligence Scale, 3rd Edition (WAIS-III), Digit Span subtest. Participants are asked to repeat digit strings that are verbally administered exactly as they hear them (digits forward) or to repeat them backwards (digits backward).
Change in processing speed | Baseline and up to day 8
  Measured by the Wechsler Adult Intelligence Scale, 3rd Edition (WAIS-III), Digit Symbol-Coding subtest. Participants are given three minutes to draw symbols as quickly and as accurately as possible according to a key code.
Change in visual memory | Baseline and up to day 8
  Measured by the Wechsler Memory Scale, 3rd Edition (WMS-III), Visual Reproduction subtest. Participants are asked to draw abstract figures from memory at different time intervals. The subtest assesses the following visual memory skills: immediate free recall, long delayed free recall and a long delayed recognition.
Change in sustained and selective attention | Baseline and up to day 8
  Measured by the Ruff 2 & 7 Selective Attention Test. The test consists of a series of 20 trials of a visual search and cancellation task. The participant detects and marks through all occurrences of the two target digits: "2" and "7." In the 10 Automatic Detection trials, the target digits are embedded among alphabetical letters that serve as distractors. In the 10 Controlled Search trials, the target digits are embedded among other numbers that serve as distractors. Correct hits and errors are counted for each trial and serve as the basis for scoring the test.
Change in working memory and attention | Baseline and up to day 8
  Measured by the Paced Auditory Serial Addition Test (PASAT). Participants are read a series of numbers at specified time intervals. The participants are instructed to add the number to the preceding number and continue adding them together until the end of the trial. Four trials with 50 items each are administered with a 30 second break in between.
Change in depression symptoms | Baseline and up to day 8
  Measured by the Beck Depression Inventory, 2nd Edition (BDI-II), which is a self-report questionnaire with 21 multiple choice items. The total score ranges from 0 to 63 with higher numbers indicating greater severity of depression symptoms.
Change in anxiety symptoms | Baseline and up to day 8
  Measured by the State Trait Anxiety Inventory (STAI), which is a self-report questionnaire with 40 questions on a 4-point likert scale. The STAI measures two types of anxiety - state and trait scores. Higher scores are positively correlated with higher levels of anxiety.

SECONDARY OUTCOMES:
Change in functional neuroimaging activation | Baseline and up to day 8
  Functional resting state sequences will be performed on the Phillips 3 tesla magnetic resonance (MR) research scanner.
Change in Symptom Score on the Sport Concussion Assessment Tool (SCAT3) | Baseline and up to day 70
  Obtained from the 22-item symptom evaluation included in the Sport Concussion Assessment Tool (SCAT3). The participant's present experience of each symptom is rated on a likert scale from 0 (none) to 6 (severe). The symptom score represents how many symptoms the participant endorses experiencing at a level greater than 0 (maximum 22 points).
Change in Symptom Severity on the Sport Concussion Assessment Tool (SCAT3) | Baseline and up to day 70
  Symptom evaluation included in the Sport Concussion Assessment Tool (SCAT3). The participant's present experience of each symptom is rated on a likert scale from 0 (none) to 6 (severe). The symptom severity represents the total summed severity ratings for all symptoms (maximum 132 points).
Change in sleep quality | Baseline and up to day 70
  Obtained from the Medical Outcomes Sleep Scale (MOS). This measure has 12 items and asks the participant to rate different aspects of their sleep experiences and sleep quality. The first two questions inquire about sleep times and the remaining questions utilize a likert scale ranging from 1 (all of the time) to 6 (none of the time).
Change in postural stability | Baseline and up to day 70
  The Balance Error Scoring System (BESS) will be used to measure postural stability, which is sensitive to deficits in balance following mild head injury. A modified version of (SCAT3) will be used. It includes three different stances, double leg, single leg, and tandem stance. A point is added for committing an error during the test interval and if the participant is unable to maintain his or her balance for more than 5 seconds, the trial is discontinued and maximum points are awarded. The total score ranges from 0 (better postural stability) to 30 (worse postural stability).
Change in depression symptoms | Baseline and up to day 70
  Measured by the Beck Depression Inventory, 2nd Edition (BDI-II), which is a self-report questionnaire with 21 multiple choice items. The total score ranges from 0 to 63 with higher numbers indicating greater severity of depression symptoms.
Change in anxiety symptoms | Baseline and up to day 70
  Measured by the State Trait Anxiety Inventory (STAI), which is a self-report questionnaire with 40 questions on a 4-point likert scale. The STAI measures two types of anxiety - state and trait scores. Higher scores are positively correlated with higher levels of anxiety.

OTHER OUTCOMES:
Change in aerobic fitness | Baseline and up to day 8
  Measured by the 3-Minute Step Test, which provides an estimate of aerobic fitness. Participants step up and down continuously on a 12-inch step for 3 minutes and the time it takes for their heart rate to return to baseline is recorded.
Change in body weight | Baseline and up to day 8
  Body weight measured in kilograms.
Minutes of physical activity outside of exercise program | Day 7 of exercise program
  Average number of minutes the participant spent engaging in physical activity outside of the exercise sessions during the one-week exercise program. This will be measured by a digital fitness monitor that will be worn 24 hours per day during the 7 day exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Russell M. Bauer, Ph.D., Principal Investigator — University of Florida; Aliyah R. Snyder, M.S., Study Director — University of Florida
Locations (1):
- University of Florida Health Science Center, Gainesville, Florida, United States

REFERENCES:
- [Background] Cassidy JD, Carroll LJ, Peloso PM, Borg J, von Holst H, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Incidence, risk factors and prevention of mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):28-60. doi: 10.1080/16501960410023732. PMID 15083870
- [Background] Barkhoudarian G, Hovda DA, Giza CC. The molecular pathophysiology of concussive brain injury. Clin Sports Med. 2011 Jan;30(1):33-48, vii-iii. doi: 10.1016/j.csm.2010.09.001. PMID 21074080
- [Background] Prins ML, Alexander D, Giza CC, Hovda DA. Repeated mild traumatic brain injury: mechanisms of cerebral vulnerability. J Neurotrauma. 2013 Jan 1;30(1):30-8. doi: 10.1089/neu.2012.2399. PMID 23025820
- [Background] Griesbach GS, Gomez-Pinilla F, Hovda DA. Time window for voluntary exercise-induced increases in hippocampal neuroplasticity molecules after traumatic brain injury is severity dependent. J Neurotrauma. 2007 Jul;24(7):1161-71. doi: 10.1089/neu.2006.0255. PMID 17610355
- [Background] Bigler ED. Neuropsychology and clinical neuroscience of persistent post-concussive syndrome. J Int Neuropsychol Soc. 2008 Jan;14(1):1-22. doi: 10.1017/S135561770808017X. PMID 18078527
- [Background] Griesbach GS, Hovda DA, Gomez-Pinilla F. Exercise-induced improvement in cognitive performance after traumatic brain injury in rats is dependent on BDNF activation. Brain Res. 2009 Sep 8;1288:105-15. doi: 10.1016/j.brainres.2009.06.045. Epub 2009 Jun 23. PMID 19555673
- [Background] Coelho FG, Gobbi S, Andreatto CA, Corazza DI, Pedroso RV, Santos-Galduroz RF. Physical exercise modulates peripheral levels of brain-derived neurotrophic factor (BDNF): a systematic review of experimental studies in the elderly. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):10-5. doi: 10.1016/j.archger.2012.06.003. Epub 2012 Jun 29. PMID 22749404
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. The DOSE study: a clinical trial to examine efficacy and dose response of exercise as treatment for depression. Control Clin Trials. 2002 Oct;23(5):584-603. doi: 10.1016/s0197-2456(02)00226-x. PMID 12392873
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Riemann BL, Guskiewicz KM. Effects of mild head injury on postural stability as measured through clinical balance testing. J Athl Train. 2000 Jan;35(1):19-25. PMID 16558603